CLINICAL TRIAL: NCT01948193
Title: Immunogenicity and Safety of Sanofi Pasteur's DTaP-IPV-Hep B-PRP-T Combined Vaccine Given at 6, 10 and 14 Weeks of Age in Infants From India Who Previously Received a Dose of Hepatitis B Vaccine at Birth
Brief Title: Study of DTaP-IPV-Hep B-PRP~T Combined Vaccine in Indian Infants Previously Given a Dose of Hepatitis B Vaccine at Birth
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: A3L33; U1111-1127-6936 (Other: WHO); CTRI/2013/09/003997 (Registry Identifier: Clinical Trial Registry India)
Record Dates: First submitted 2013-09-18; First posted 2013-09-23 (Estimated); Results first posted 2015-09-25 (Estimated); Last update posted 2015-10-20 (Estimated); Status verified 2015-09

CONDITIONS: Diphtheria; Tetanus; Whooping Cough; Hepatitis B; Poliomyelitis; Invasive Hib Infections
Keywords: Diphtheria; Tetanus; Whooping Cough; Hepatitis B; Poliomyelitis; DTaP IPV-Hep B-PRP~T combined vaccine (Hexaxim™)
MeSH Terms: conditions — Diphtheria; Tetanus; Whooping Cough; Hepatitis B; Poliomyelitis | interventions — DTaP-IPV-HB-PRP-T vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Study Group (Experimental): Participants will receive Sanofi Pasteur's DTaP-IPV-Hep B-PRP~T combined vaccine (investigational vaccine) at 6, 10 and 14 weeks of age.
  Interventions: Biological: Hexaxim™: DTaP-IPV-Hep B-PRP~T combined vaccine

INTERVENTIONS:
Biological: Hexaxim™: DTaP-IPV-Hep B-PRP~T combined vaccine — 0.5 mL, Intramuscular
  Other Names: Hexaxim™

SUMMARY:
The purpose of this study is to describe the immunogenicity and safety of a novel DTaP- IPV- Hep B-PRT~T fully liquid combined hexavalent vaccine (Hexaxim™) administered at 6, 10 and 14 weeks of age in infants born to mothers documented to be serum anti-hepatitis B surface antigen (HBsAg) serology negative in India.

Primary Objective:

* To evaluate the immunogenicity of the study vaccine in terms of seroprotection [diphtheria toxoid, tetanus toxoid, poliovirus types 1, 2 and 3, Haemophilus influenzae type b (Hib) polysaccharide (PRP), hepatitis B (Hep B)] and vaccine response for pertussis antigens [pertussis toxoid (PT) and filamentous haemagglutinin (FHA)] one month after the third dose.

Secondary Objectives:

* To further describe the immunogenicity of the study vaccine, before the first dose and one month after the third dose.
* To describe the safety after each and any doses of the study vaccine.

DETAILED DESCRIPTION:
All participants will receive a total 4 doses of Hep B, i.e. one dose of Hep B monovalent vaccine given at birth followed by 3 doses of Sanofi Pasteur's hexavalent vaccine given at 6, 10 and 14 weeks of age in the context of the study. Participants and parents will attend four clinic visits; the expected participation in the study is approximately 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 42-56 days (6 to 8 weeks) on the day of inclusion
* Born at full term of pregnancy (≥37 weeks) and with a birth weight ≥2.5 kg
* Informed consent form signed by the parent(s) or any other legally acceptable representative
* Subject and parent/legally acceptable representative are able to attend all scheduled visits and to comply with all trial procedures
* Born to known hepatitis B surface antigen (HBsAg) seronegative mother (documented laboratory result of HBsAg assay from maternal blood sample performed during last trimester of pregnancy available)
* Have received one documented dose of Hep B vaccine and oral poliovirus vaccine (OPV) from birth as per national recommendations.

Exclusion Criteria:

* Participation in another clinical trial in the 4 weeks preceding the trial inclusion or planned participation during the present trial period in another clinical trial investigating a vaccine, drug, medical device, or medical procedure
* Receipt of any vaccine in the 4 weeks preceding the first trial vaccination (except Bacillus Calmette-Guerin [BCG] vaccine) or planned receipt of any other vaccine within the period from 8 days before to 8 days after each subsequent trial vaccination
* Previous vaccination against the diphtheria, tetanus, pertussis, poliomyelitis (expect the birth dose of OPV as per national recommendations) and hepatitis B (except the birth dose of Hep B vaccine) diseases or Hib infection with the trial vaccine or another vaccine
* Past or current receipt of immune globulins, blood or blood-derived products or planned administration during the trial
* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy, such as anti-cancer chemotherapy or radiation therapy since birth; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks since birth)
* History of diphtheria, tetanus, pertussis, poliomyelitis, hepatitis B, or Hib infections (confirmed either clinically, serologically or microbiologically)
* Known personal or maternal history of Human Immunodeficiency Virus (HIV) or hepatitis C seropositivity
* Known systemic hypersensitivity to any of the vaccine components, or history of a life-threatening reaction to the trial vaccine or a vaccine containing the same substances
* Known thrombocytopenia, as reported by the parent/legally acceptable representative
* Bleeding disorder, or receipt of anticoagulants in the 3 weeks preceding inclusion, contraindicating intramuscular vaccination
* In an emergency setting, or hospitalized involuntarily
* Chronic illness that, in the opinion of the investigator, is at a stage where it might interfere with trial conduct or completion
* Moderate or severe acute illness/infection (according to investigator judgment) on the day of vaccination or febrile illness (axillary temperature ≥38°C) on the day of inclusion (a prospective subject should not be included in the study until the condition has resolved or the febrile event has subsided)
* Identified as a natural or adopted child of the Investigator, relatives or employee with direct involvement in the proposed study
* History of seizures.

Ages: 6 Weeks to 8 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 177 (Actual)
Dates: Start 2014-02; Primary Completion 2014-12 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur SA
Locations (2):
- India (2):
  - Ludhiana, Punjab
  - Pune

REFERENCES:
- See also: Related Info — http://www.sanofipasteur.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study participants were enrolled from 19 February 2014 to 30 June 2014 at 2 clinical sites in India.
Pre-assignment Details: A total of 177 participants who met all of the inclusion criteria and none of the exclusion criteria were enrolled and vaccinated.
Groups:
- All Infants: Infants aged 6 to 8 weeks received 3 injections of Sanofi Pasteur's DTaP IPV HB PRP T combined vaccine at 6, 10 and 14 weeks of age following a documented dose of a commercial oral poliovirus vaccine and recombinant Hepatitis B monovalent vaccine at birth.
Period: Overall Study
Arm/Group | All Infants
Started | 177
Completed | 168
Not Completed | 9
Not completed — Serious event | 2
Not completed — Lost to Follow-up | 7

BASELINE CHARACTERISTICS:
Groups:
- All Infants: Infants aged 6 to 8 weeks received 3 injections of Sanofi Pasteur's DTaP-IPV-HB-PRP-T combined vaccine at 6, 10 and 14 weeks of age following a documented dose of a commercial oral poliovirus vaccine and recombinant Hepatitis B monovalent vaccine at birth.
Arm/Group | All Infants
Number analyzed (Participants) | 177
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 177
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: Weeks] | 6.9 (0.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 78
  Male | 99
Region of Enrollment [Number; unit: Participants]
  India | 177

OUTCOME MEASURES:

1. Secondary Outcome: Percentage of Participants With Seroprotection Before and After Vaccinations With Sanofi Pasteur's DTaP-IPV-HB-PRP-T Combined Vaccine Following a Documented Dose of a Commercial Oral Poliovirus Vaccine and Recombinant Hep B Monovalent Vaccine at Birth
Description: Diphtheria antibodies were measured by a toxin neutralization test, tetanus antibodies by an enzyme-linked immunosorbent assay (ELISA), Haemophilus influenzae type b polysaccharide (PRP) antibodies by Farr type radioimmunoassay, poliovirus 1, 2, and 3 antibodies by a neutralization assay, and Hepatitis B (Hep B) antibodies were measured by VITROS ECi/ECiQ Immunodiagnostic System.
  Description of seroprotection: Diphtheria and Tetanus antibody concentrations ≥0.01 International Units (IU)/mL; Poliovirus 1, 2, and 3 titers ≥8 (1/dilution); Hep B concentrations ≥10 mIU/mL, and PRP ≥0.15 µg/mL.
Time Frame: Pre-dose 1 to one month post-dose 3
Population: Seroprotection was assessed in the Per-protocol Analysis Set.
Measure: Number; unit: Percentage of participants
Arm/Group | All Infants
Number analyzed (Participants) | 156
Percentage of participants
  Anti-Diphtheria; Pre-dose, 1 ≥0.01 (N=152) | 67.1
  Anti-Diphtheria; Pre-dose 1, ≥0.1 (N=152) | 15.8
  Anti-Diphtheria; Post-dose 3; ≥0.01, (N=135) | 99.3
  Anti-Diphtheria; Post-dose 3; ≥0.1 (N=135) | 49.6
  Anti-Diphtheria; Post-dose 3, ≥1.0 (N=135) | 5.2
  Anti-Tetanus; Post-dose 3, ≥0.01 (N=134) | 100.0
  Anti-Tetanus; Post-dose 3, ≥0.1 (N=134) | 100.0
  Anti-Tetanus; Post-dose 3, ≥1.0 (N=134) | 84.3
  Anti-Polio 1; Post-dose 3 (N=145) | 100.0
  Anti-Polio 2; Post-dose 3 (N=146) | 100.0
  Anti-Polio 3; Post-dose 3 (N=144) | 100.0
  Anti-Hep B; Pre-dose 1, ≥10 (N=152) | 13.2
  Anti-Hep B; Post-dose 3, ≥10 (N=152) | 100.0
  Anti-Hep B; Post-dose 3, ≥100 (N=152) | 99.3
  Anti-PRP; Post-dose 3, ≥0.15 (N=156) | 100.0
  Anti-PRP; Post-dose 3, ≥1.0 (N=156) | 93.6

2. Primary Outcome: Percentage of Participants With Seroprotection After Vaccinations With Sanofi Pasteur's DTaP-IPV-HB-PRP-T Combined Vaccine Following a Documented Dose of a Commercial Oral Poliovirus Vaccine and Recombinant Hep B Monovalent Vaccine at Birth
Description: as for outcome 1
Time Frame: Pre-dose 1 to one month post-dose 3
Population: Seroprotection was assessed in the Per-protocol Analysis Set.
Measure: Number; unit: Percentage of participants
Arm/Group | All Infants
Number analyzed (Participants) | 156
Percentage of participants
  Anti-Diphtheria; Post-dose 3; ≥0.01, (N=135) | 99.3
  Anti-Tetanus; Post-dose 3, ≥0.01 (N=134) | 100
  Anti-Polio 1; Post-dose 3 (N=145) | 100
  Anti-Polio 2; Post-dose 3 (N=146) | 100
  Anti-Polio 3; Post-dose 3 (N=144) | 100
  Anti-Hep B; Post-dose 3, ≥10 (N=152) | 100
  Anti-PRP; Post-dose 3, ≥0.15 (N=156) | 100

3. Secondary Outcome: Geometric Mean Titers of Antibodies Against Vaccine Antigens After Vaccinations With Sanofi Pasteur's DTaP-IPV-HB-PRP-T Combined Vaccine After a Documented Dose of an Oral Poliovirus Vaccine and Recombinant Hep B Monovalent Vaccine at Birth
Description: Diphtheria antibodies were measured by a toxin neutralization test, tetanus, PT, and FHA antibodies by an ELISA, PRP antibodies by a Farr type radioimmunoassay, poliovirus 1, 2, and 3 antibodies by a neutralization assay, and Hep B antibodies were measured by VITROS ECi/ECiQ Immunodiagnostic System.
Time Frame: Pre-dose 1 to one month post-dose 3
Population: Geometric mean titers were assessed in the Per-protocol Analysis Set.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | All Infants
Number analyzed (Participants) | 156
Titers
  Anti-Diphtheria; Pre-dose 1 (N=152) | 0.019 [0.015 to 0.025]
  Anti-Diphtheria; Post-dose 3 (N=135) | 0.120 [0.099 to 0.146]
  Anti-Tetanus; Post-dose 3 (N=134) | 1.95 [1.75 to 2.17]
  Anti-PT; Pre-dose 1 (N=147) | 3.84 [3.00 to 4.91]
  Anti-PT; Post-dose 3 (N=155) | 191 [173 to 210]
  Anti-FHA; Pre-dose 1 (N=151) | 6.17 [5.10 to 7.48]
  Anti-FHA; Post-dose 3 (N=152) | 226 [208 to 247]
  Anti-Polio 1; Post-dose 3 (N=145) | 1124 [861 to 1468]
  Anti-Polio 2; Post-dose 3 (N=146) | 1401 [1108 to 1771]
  Anti-Polio 3; Post-dose 3 (N=144) | 2019 [1672 to 2437]
  Anti-Hep B; Pre-dose 1 (N=152) | 3.78 [3.23 to 4.43]
  Anti-Hep B; Post-dose 3 (N=152) | 2491 [2073 to 2995]
  Anti-PRP; Post-dose 3 (N=156) | 7.86 [6.35 to 9.73]

4. Secondary Outcome: Geometric Mean Titer Ratios of Antibodies Against Vaccine Antigens After Vaccinations With Sanofi Pasteur's DTaP-IPV-HB-PRP-T Combined Vaccine After a Documented Dose of Oral Poliovirus Vaccine and Recombinant Hep B Monovalent Vaccine at Birth
Description: Diphtheria antibodies were measured by a toxin neutralization test, PT and FHA antibodies by an ELISA, and Hep B antibodies were measured by VITROS ECi/ECiQ Immunodiagnostic System.
Time Frame: Pre-dose 1 to one month post-dose 3
Population: Geometric mean titer ratios were assessed in the Per-protocol Analysis Set.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer ratio
Arm/Group | All Infants
Number analyzed (Participants) | 156
Titer ratio
  Anti-Diphtheria (N=131) | 5.85 [3.93 to 8.72]
  Anti-PT (N=146) | 50.7 [37.3 to 69.0]
  Anti-FHA (N=147) | 36.6 [28.6 to 46.8]
  Anti-Hep B (N=149) | 686 [542 to 870]

5. Secondary Outcome: Percentage of Participants Reporting Solicited Injection-site or Systemic Reaction After Each Vaccination With Sanofi Pasteur's DTaP-IPV-HB-PRP-T Combined Vaccine Following a Documented Dose of Oral Poliovirus and Recombinant Hep B Vaccine at Birth
Description: Injection-site reactions: Tenderness, Erythema, and Swelling. Systemic reactions: Fever, Vomiting, Crying abnormal, Drowsiness, Appetite lost, and Irritability. Grade 3 Injection site reactions: Tenderness, Cries when injected limb is moved, or reduced movement of injected limb; Erythema and Swelling, ≥50 mm. Grade 3 Systemic reactions: Fever, >39.5°C or >103.1°F; Vomiting, ≥6 episodes/24 hours or requires parenteral hydration; Crying abnormal, >3 hours; Drowsiness, Sleeping most of the time/difficult to wake up; Appetite lost, Refuses ≥3 or most feeds/meals; Irritability, Inconsolable.
Time Frame: Within 7 days after each vaccine injection
Population: Solicited injection-site and systemic reactions were assessed in the Safety Analysis Set.
Measure: Number; unit: Percentage of participants
Arm/Group | All Infants
Number analyzed (Participants) | 177
Percentage of participants
  Any Injection-site Tenderness; Post Inj. 1 (N=174) | 19.0
  Grade 3 Inj. site Tenderness; Post Inj 1 (N=174) | 2.3
  Any Injection-site Erythema; Post Inj. 1 (N=174) | 4.6
  Grade 3 Inj. site Erythema; Post Inj. 1 (N=174) | 0.0
  Any Injection-site Swelling; Post Inj. 1 (N=174) | 10.3
  Grade 3 Inj. site Swelling; Post Inj. 1 (N=174) | 0.0
  Any Injection-site Tenderness; Post Inj. 2 (N=174) | 13.8
  Grade 3 Inj.-site Tenderness; Post Inj. 2 (N=174) | 1.1
  Any Injection-site Erythema; Post Inj. 2 (N=174) | 3.4
  Grade 3 Inj. site Erythema; Post Inj. 2 (N=174) | 0.0
  Any Injection-site Swelling; Post Inj. 2 (N=174) | 3.4
  Grade 3 Inj. site Swelling; Post Inj. 2 (N=174) | 0.0
  Any Injection-site Tenderness; Post Inj. 3 (N=168) | 11.9
  Grade 3 Inj. site Tenderness; Post Inj. 3 (N=168) | 0.0
  Any Injection-site Erythema; Post Inj. 3 (N=168) | 0.6
  Grade 3 Inj. site Erythema; Post Inj. 3 (N=168) | 0.0
  Any Injection-site Swelling; Post Inj. 3 (N=168) | 6.5
  Grade 3 Inj. site Swelling; Post Inj. 3 (N=168) | 0.0
  Any Fever; Post-injection 1 (N=174) | 7.5
  Grade 3 Fever; Post-injection 1 (N=174) | 0.0
  Any Vomiting; Post-injection 1 (N=174) | 9.8
  Grade 3 Vomiting; Post-injection 1 (N=174) | 0.0
  Any Crying abnormal; Post-injection 1 (N=174) | 16.1
  Grade 3 Crying abnormal; Post-injection 1 (N=174) | 1.1
  Any Drowsiness; Post injection 1 (N=174) | 9.8
  Grade 3 Drowsiness; Post Inj. 1 (N=174) | 1.1
  Any Appetite lost; Post Inj. 1 (N=174) | 6.9
  Grade 3 Appetite lost; Post Inj. 1 (N=174) | 0.0
  Any Irritability; Post Inj. 1 (N=174) | 22.4
  Grade 3 Irritability; Post Inj. 1 (N=174) | 0.6
  Any Fever; Post Inj. 2 (N=174) | 8.6
  Grade 3 Fever; Post Inj. 2 (N=174) | 0.0
  Any Vomiting; Post Inj. 2 (N=174) | 3.4
  Grade 3 Vomiting; Post Inj. 2 (N=174) | 0.0
  Any Crying abnormal; Post Inj. 2 (N=174) | 9.8
  Grade 3 Crying abnormal; Post Inj. 2 (N=174) | 0.0
  Any Drowsiness; Post Inj. 2 (N=174) | 3.4
  Grade 3 Drowsiness; Post Inj. 2 (N=174) | 0.0
  Any Appetite lost; Post Inj. 2 (N=174) | 3.4
  Grade 3 Appetite lost; Post Inj. 2 (N=174) | 0.0
  Any Irritability; Post Inj. 2 (N=174) | 16.7
  Grade 3 Irritability; Post Inj. 2 (N=174) | 0.0
  Any Fever; Post Inj. 3 (N=168) | 7.1
  Grade 3 Fever; Post Inj. 3 (N=168) | 0.0
  Any Vomiting; Post Inj. 3 (N=168) | 3.0
  Grade 3 Vomiting; Post Inj. 3 (N=168) | 0.0
  Any Crying abnormal; Post Inj. 3 (N=168) | 7.7
  Grade 3 Crying abnormal; Post Inj. 3 (N=168) | 0.0
  Any Drowsiness; Post Inj. 3 (N=168) | 3.0
  Grade 3 Drowsiness; Post Inj. 3 (N=168) | 0.0
  Any Appetite lost; Post Inj. 3 (N=168) | 3.0
  Grade 3 Appetite lost; Post Inj. 3 (N=168) | 0.0
  Any Irritability; Post Inj. 3 (N=168) | 12.5
  Grade 3 Irritability; Post Inj. 3 (N=168) | 0.0

6. Primary Outcome: Percentage of Participants With Vaccine Response After Vaccinations With Sanofi Pasteur's DTaP-IPV-HB-PRP-T Combined Vaccine Following a Documented Dose of a Commercial Oral Poliovirus Vaccine and Recombinant Hep B Monovalent Vaccine at Birth
Description: Anti-pertussis toxin (PT) and anti-filamentous hemagglutinin (FHA) antibodies were measured with an ELISA. Vaccine response was defined as percentage of participants with post-dose 3 anti-PT and anti-FHA antibody concentrations in ELISA units (EU)/mL ≥ 4 x Lower Limit of Quantification (LLOQ) if pre-vaccination concentration was < 4 x LLOQ or ≥ pre-vaccination concentration if pre-vaccination concentrations ≥ 4 x LLOQ.
Time Frame: Pre-dose 1 to one month post-dose 3
Population: Vaccine response was assessed in the Per-protocol Analysis Set.
Measure: Number; unit: Percentage of participants
Arm/Group | All Infants
Number analyzed (Participants) | 156
Percentage of participants
  Anti-PT; Pre-dose 1 (N=147) | 59.9
  Anti-PT; Vaccine response (N=146) | 93.8
  Anti-PT; ≥4-fold increase (N=146) | 88.4
  Anti-FHA; Pre-dose 1 (N=151) | 88.7
  Anti-FHA; Vaccine response (N=147) | 99.3
  Anti-FHA; ≥4-fold increase (N=147) | 90.5

ADVERSE EVENTS:
Time Frame: Adverse event data were collected following first vaccination up to Day 30 post-dose 3.
Arm/Group | All Infants
Serious Adverse Events (participants affected / at risk) | 3/177
Other Adverse Events (participants affected / at risk) | 39/177
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Infants (N=177)
Death unexplained (General disorders) | 1 (1)
Bronchopneumonia (Infections and infestations) | 1 (1)
Septic shock (Infections and infestations) | 1 (1)
Epilepsy (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5.00% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | All Infants (N=177)
Diarrhoea (Gastrointestinal disorders) | 9 (9)
Upper respiratory tract infection (Infections and infestations) | 21 (24)
Injection site Tenderness (General disorders) | 33/174 (33)
Injection site Erythema (General disorders) | 8/174 (8)
Injection site Swelling (General disorders) | 18/174 (18)
Fever (General disorders) | 15/174 (15)
Vomiting (Gastrointestinal disorders) | 17/174 (17)
Crying abnormal (Psychiatric disorders) | 28/174 (28)
Drowsiness (Nervous system disorders) | 17/174 (17)
Appetite lost (Metabolism and nutrition disorders) | 12/174 (12)
Irritability (Psychiatric disorders) | 39/174 (39)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications